CLINICAL TRIAL: NCT07180082
Title: Continuous or Intermittent Pyrotinib for HER2-positive Advanced Breast Cancer: a Prospective, Randomized, Controlled, Multicentre Clinical Trial
Brief Title: Continuous or Intermittent Pyrotinib for HER2-positive Advanced Breast Cancer
Acronym: CORIN-PYRA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wenjin Yin (Other)
Responsible Party: Sponsor-Investigator, Wenjin Yin, Deputy Chief of Breast Surgery Department, RenJi Hospital
Organization: RenJi Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY2025-118-A
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — pyrotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent pyrotinib (Experimental): Intermittent use of pyrotinib, 14 days on and 7 days of, every 21 days
  Interventions: Drug: Pyrotinib
- Continuous pyroitnib (Active Comparator): oral pyrotinib qd
  Interventions: Drug: Pyrotinib

INTERVENTIONS:
Drug: Pyrotinib — anti-HER2 tyrosine kinase inhibitor

SUMMARY:
This is a prospective, randomised, controlled, multicentre study to evaluate the efficacy and safety of continuous versus intermittent pyrotinib therapy in patients with human epidermal growth factor receptor (HER2)-positive advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years old
* Pathologically confirmed advanced or locally advanced breast cancer not amenable to curative surgery
* Pathologically confirmed HER2+ at least once for either primary or metastatic lesion
* Previously treated with any number of lines for advanced disease and eligible for a pyrotinib-containing regimen at the discretion of physician
* At least one measurable lesion or bone-only disease (osteolytic or mixed) according to RECIST v1.1
* ECOG 0-1
* Adequate organ function

Exclusion Criteria:

* During pregnancy and lactation
* Difficulties with pyrotinib administration or absorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | From the date of starting pyrotinib to the date of confirmed CR or PR (up to approximately 1 years)
  ORR is the percentage of subjects with complete remission (CR) or partial remission (PR) as the best response during the period from the beginning of the treatment to the progression of the disease or the completion of therapy (CR+PR)/Analysis of the total number of people. Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) was used to assess the objective tumor response.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From the date of starting pyrotinib to the date of first documentation of disease progression or death from any cause (up to approximately 1 year)
  PFS is defined as the time from the date of starting maintenance therapy to the date of disease progression or death from any cause, whichever occurs first.
Adverse events | From the date of starting pyrotinib to the end of the treatment (up to approximately 1 year)
  Adverse events during maintenance therapy will be assessed according to the NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Wenjin Yin, M.D., Principal Investigator — Renji Hospital,School of Medicine, Shanghai Jiaotong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No